CLINICAL TRIAL: NCT01392872
Title: Evaluation of Cognitive Disability and Quality of Life of Patients Suffering From Multiple Scleroses and Treat With Immunosuppressant
Brief Title: Cognitive Disability and Quality of Life of Patients Suffering From Multiple Sclerosis and Treatment With Immunosuppressant
Acronym: CoQualSEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Bordeaux (Other); University Hospital, Caen (Other); University Hospital, Marseille (Other); Dr Remy MORELLO - CHU de Caen (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHU-0094
Record Dates: First submitted 2011-05-05; First posted 2011-07-13 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2016-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Immunosuppressant; Quality of life; Cognitive function; Relapsing Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Neuropsychological Tests

ARMS (1):
- sclerosis (Other)
  Interventions: Other: Neuropsychological assessment

INTERVENTIONS:
Other: Neuropsychological assessment — This study will evaluate the impact of these treatments on cognitive disabilities, tiredness state, emotion and quality of life in general, on a lengthened period.

SUMMARY:
Multiple Sclerosis is the first cause of neurological handicap in France. The importance of cognitive disabilities, their evaluation and their impact on patients' life have only been comprehended recently. Immunosuppressants represent new treatments in Multiple Sclerosis (MS) but imply a lot of constraints. This study will evaluate the impact of these treatments on cognitive disabilities, tiredness state, emotion and quality of life in general, on a lengthened period.

DETAILED DESCRIPTION:
Multiple Sclerosis is the first cause of neurological handicap in France. The importance of cognitive disabilities, their evaluation and their impact on patients' life have only been comprehended recently. Immunosuppressants represent new treatments in MS but imply a lot of constraints. This study will evaluate the impact of these treatments on cognitive disabilities, tiredness state, emotion and quality of life in general, on a lengthened period.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Relapsing MS since at least 6 months and less than 10 years
* Neurological state stable since at least 1 month
* Moderate Handicap (EDSS ≤ 5,5)

Exclusion Criteria:

* Secondary Progressive MS
* Patient having an attack
* Patient having experienced en MS relapse or recovered systemic corticosteroid in the previous 1 month
* Depressive patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2009-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evolution of the quality of life of patients diagnosed with relapsing MS and starting a treatment with immunosuppressant | on a 36 months period

SECONDARY OUTCOMES:
Analysis of variance for repeated measurement | 15 to 30 days before the beginning of treatment, after 36 months
Selective Reminding Test (SRT) | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 18 and 36 months
Delayed recall of SRT | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 18 and 36 months
Visuo-spatial span | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 18 and 36 months
Digit span | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 18 and 36 months
Reverse span | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 18 and 36 months
Stroop test | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 18 and 36 months
• Tiredness (EMIF SEP scale): Analysis of variance for repeated measurement | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 6,12,18 and 36 months
• Physical function (9HPT, 8 meter walk) : Analysis of variance for repeated measurement | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 6,12,18 and 36 months
Disability (EDSS) : Analysis of variance for repeated measurement | 15 to 30 days before the beginning of treatment, 1st day of treatment, after 6,12,18 and 36 months
• Psychological disorder (Beck depression inventory, COVI scale, Depressive scale) : Analysis of variance for repeated measurement | 15 to 30 days before the beginning of treatment, 1st day of the treatment, after 6,12,18 and 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CLAVELOU, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Planche V, Moisset X, Morello R, Dumont E, Gibelin M, Charre-Morin J, Saubusse A, Mondou A, Reuter F, Defer G, Pelletier J, Brochet B, Clavelou P. Improvement of quality of life and its relationship with neuropsychiatric outcomes in patients with multiple sclerosis starting treatment with natalizumab: A 3-year follow-up multicentric study. J Neurol Sci. 2017 Nov 15;382:148-154. doi: 10.1016/j.jns.2017.10.008. Epub 2017 Oct 6. PMID 29111011